CLINICAL TRIAL: NCT01433744
Title: Short-term Changes on C-Reactive Protein (CRP) Levels After Non-surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of Maringá (Other)
Responsible Party: Principal Investigator, André Barbisan de Souza, DDS, State University of Maringá
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5209/2009
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Periodontitis; Atherosclerotic Cardiovascular Disease
Keywords: C-Reactive protein; risk
MeSH Terms: conditions — Chronic Periodontitis; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chronic periodontal disease (Experimental): C-reactive protein levels assesments and periodontal treatment
  Interventions: Procedure: Non-surgical periodontal treatment
- Periodontally healthy (No Intervention)

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Patients included in the test group were submitted to a non-surgical periodontal treatment protocol, which consisted of oral hygiene orientation and motivation followed by mechanical plaque control involving scaling and root planning using Gracey curets (Hu-Friedy Manufacturing, Chicago, IL, USA) and ultrasonic instrumentation (Cavitron Ultrasonics, Long Island City, NY, USA), under local anesthesia (Mepivacaine 2% with epinephrine 1:100000). The treatment was performed in one or two sessions depending on the extension of the patient's periodontal condition. Patients that presented teeth unreasonable to treat due to advanced periodontitis, or any other condition were extracted under local anesthesia.
  Arms: Chronic periodontal disease

SUMMARY:
The hypotheses tested were that levels of C-Reactive Protein (CRP) would be higher in patients with chronic periodontitis in comparison with those without periodontal disease and that the non-surgical periodontal treatment would decrease levels of CRP in patients with chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

Patients should have ≥ 20 teeth present; (ii) absence of oral soft tissue lesions; (iii) have ≤ 3 carious lesions in all teeth. In addition, to be included in the Test group the subject had to present chronic periodontitis (involvement of at least 5 teeth with at least one site presenting probing depth (PD) ≥ 5 mm and clinical attachment loss (CAL) ≥ 3 mm) while to be included in the Control group the patient had to exhibit periodontal healthy (bleeding on probing (BOP) < 30% of the sites and absence of any PD > 4mm associated with BOP).

Exclusion Criteria:

(i) periodontal disease treatment in the previous six months; (ii) aged less than 35 years; (iii) systemic conditions such as history of CVD or any other chronic or immunologic diseases and the use of related drugs in the previous six months; (iv) smokers or former smokers; (v) pregnant or lactating women; (vi) hypertension (>140 systolic and > 90 diastolic mmHg); (vii) obesity (Body Mass Index (BMI) ≥ 30 kg/m²); (viii) levels of HDL-cholesterol > 35.0 mg/dL (ix) levels of LDL-cholesterol < 160.0 mg/dL (x)levels of triglycerides < 400.0 mg/dL and (xi) levels of glucose levels < 100 mg/dL.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
C-Reactive Protein levels | Baseline and 60 days after treatment

SECONDARY OUTCOMES:
The effect of non-surgical periodontal treatment on patients with chronic periodontitis | Baseline and re-evaluation 60 days after the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Departament of Dentistry of State University of Maringá, Maringá, Paraná, Brazil